CLINICAL TRIAL: NCT01744678
Title: Experimental Trial of Fatigue Countermeasure Program in Operational Flight Controllers
Brief Title: Fatigue Countermeasure Program in Operational Flight Controllers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Chief, Division of Sleep Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NNX10AF47G
Record Dates: First submitted 2012-10-11; First posted 2012-12-07 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Access to experimental break room (Experimental): Subjects will visit the experimental break room 4 times per Orbit 1 shift:
  * first, prior to the beginning of the work shift
  * second, during an operationally feasible 20-min break during the 1st half of the work shift
  * third, once during an operationally feasible 20-min break during the 2nd half of the work shift
  * fourth, immediately after the end of the work shift
  In the break room, subjects will be passively exposed to blue-wavelength enriched ceiling lights during all four visits for each work shift.
  Also in the break room, subjects will perform 10-minutes of mild exercise during the first three visits to the break room during each work shift.
  Interventions: Behavioral: blue-wavelength enriched ceiling light; Behavioral: mild exercise

INTERVENTIONS:
Behavioral: blue-wavelength enriched ceiling light — Subjects will be in the experimental break room for four 20-minute periods for each Orbit 1 work shift.
  Other Names: Sylvania Fluorescent Octron FO32/SKYWHITE/XP/ECO 8000K
Behavioral: mild exercise — Subjects will be asked to achieve 65% of maximum heart rate on either a treadmill or exercise cycle for 10-minutes, three times during each Orbit 1 work shift.
  Other Names: ICON Health and Fitness Pro2000 Treadmill PFTL13011; ICON Health and Fitness 290SPX Bike PFEX02909

SUMMARY:
The purpose of this study is to validate the acceptability, operational feasibility and efficacy of a combined fatigue countermeasure comprised of shorter-wavelength light and exercise during operational Orbit 1 night shifts to improve alertness and performance of flight mission controllers.

Specifically, the investigators will:

1. Feasibility. Test the feasibility of developing a break room containing fatigue countermeasures (shorter-wavelength light and exercise equipment) to be used by flight mission controllers during Orbit 1 night shifts, and the feasibility to schedule regular breaks during the Orbit 1 shift so that flight mission controllers have the opportunity to use the fatigue countermeasures break room.
2. Acceptability. Test the acceptability of the use of the fatigue countermeasures break room evaluating when and how the room is used by flight mission controllers, as measured on End-of-Shift Productivity Questionnaire.
3. Test the hypothesis that alertness and performance will be impaired in flight mission controllers during Orbit 1 operational night shifts as compared to flight mission controllers working a non-console day shift.
4. Test the hypothesis that alertness and performance of flight mission controllers who exercise and are exposed to shorter wavelength light during the Orbit 1 night shift will be significantly more alert and have better mood, performance (e.g., less Psychomotor Vigilance Task (PVT) lapses, increased productivity) than those same mission controllers working Orbit 1 night shifts without exposure to the shorter wavelength light and exercise.
5. Test the acceptability, operational feasibility and efficacy of implementing an anonymous sleep disorders screening for flight controllers, evaluated by number of visitors to the screening web site and the number of completed assessments.

DETAILED DESCRIPTION:
Each participant will have three data collection periods. Each data collection period will last one shift rotation (5 -7 days): One 5-shift or 7-shift block of Orbit 1 night shifts on console with access to photic and exercise countermeasures, a second 5-shift or 7-shift block of Orbit 1 night shifts on console with no access to countermeasures, and a third 5-shift block of daytime office work off console. We will be measuring sleep via a wrist worn activity measuring device and compliance of exercise intervention via a small, commercially available heart monitor worn around the chest underneath clothing. The activity device will be worn continuously and the heart monitor will be worn on shift. These devices will be downloaded at the end of each block of shifts. Subjects will complete a short baseline questionnaire once at the beginning of the study. Subjective alertness will be assessed with the Karolinska Sleepiness Scale (KSS), performance testing will occur regularly and 'end of shift' questionnaires will be completed at the end of each shift. Drowsiness will be measured on the commute to and from work with the Optalert.

ELIGIBILITY:
Inclusion Criteria:

* Must be current Johnson Space Center International Space Station Flight Controller or Flight Director cleared to sit console for Orbit 1 work shift
* Work schedule must meet both study needs and National Aeronautics and Space Administration (NASA) scheduling operational constraints

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Alertness/Fatigue as measured by Psychomotor Vigilance Task and Visual Analog Scales | Three weeks.
  Average slowest 10% reaction times by condition (day shift, overnight control, overnight intervention), across time within shifts (pre-shift, first half, second half, post-shift), and across consecutive shifts (shifts 1, 2, 3, 4, 5)

SECONDARY OUTCOMES:
Sleep duration as measured by wrist actigraphy | Three weeks.
  Average hours of sleep per 24hr day by condition (day shift, overnight control, overnight intervention)
Sleep duration as captured in sleep/work logs | Three weeks.
  Average hours of sleep per 24hr day by condition (day shift, overnight control, overnight intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, PhD, MD, Principal Investigator — Brigham and Women's Hospital / Harvard Medical School; Laura K Barger, PhD, Study Director — Brigham and Women's Hospital / Harvard Medical School
Locations (1):
- Johnson Space Center, Houston, Texas, United States